CLINICAL TRIAL: NCT02947958
Title: Evaluation of the Effectiveness of the Use of Teleconsultation in Qualifying Counter-reference Between Tertiary and Primary Care for Patients With Benign Prostatic Hyperplasia: Randomized Clinical Trial of Noninferiority
Brief Title: Teleconsultation in Counter-reference Between Tertiary and Primary Care for Patients With Benign Prostatic Hyperplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 28976614000005327
Record Dates: First submitted 2016-10-20; First posted 2016-10-28 (Estimated); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Prostatic Hyperplasia
Keywords: teleconsultation; urology; primary care; tertiary care
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Remote Consultation; Hospitals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Teleconsultation (Experimental): Tele consultation (experimental) - after the randomization the patient is guided to seek primary care under teleconsultation supervision to keep his treatment. One year later the patient's symptoms are reassessed in a medical consultation.
  Interventions: Other: Teleconsultation
- Hospital (Active Comparator): Hospital (control) - after the randomization the patient is guided to keep his treatment in the tertiary care as usual. One year later the patient's symptoms are reassessed in a medical consultation.
  Interventions: Other: Hospital (control)

INTERVENTIONS:
Other: Teleconsultation — Teleconsultation - the teleconsultation usage in chronic diseases, such as benign hyperplasia, seems to be a promising scenario. Once the patient symptoms are evaluated and diagnosed as a stable disease he is able to keep his treatment annually. In a way to do not overload de tertiary system, such monitoring could be done under a teleconsultation with a urological supervision in the primary care.
  Arms: Teleconsultation
Other: Hospital (control) — The patient will keep his usual care at the tertiary care.
  Arms: Hospital

SUMMARY:
To evaluate the effectiveness of the use of teleconsultation in qualifying counter-reference between tertiary and primary care for patients with stable benign prostatic hyperplasia (BPH) symptoms.

DETAILED DESCRIPTION:
The effectiveness of the use of teleconsultation will be evaluated by the initial international prostate symptom score (IPSS) in patients randomized to the standard monitoring (tertiary hospital) and teleconsultation monitoring (primary care) and after twelve months.

ELIGIBILITY:
Inclusion Criteria:

* males, over forty years, with clinical diagnosis or imaging diagnosis of benign prostate hyperplasia (ultrasonography, computed tomography, magnetic resonance imaging) with stable low urinary tract symptoms and International Prostate Symptom Score lower or equal to 25 points followed at tertiary care clinic.

Exclusion Criteria:

* low urinary tract symptoms and International Prostate Symptom Score over to 25 points, inadequate clinical treatment response, surgical treatment indication, suspicion of prostate malignancy or urethra stricture or neurogenic bladder and illiterates.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline Low Urinary Tract Symptoms (LUTS) | 12 months
  Low urinary tract symptoms are assessed through International Prostate Score System (IPSS) which includes seven main important symptoms of benign prostate hyperplasia, validated to portuguese. Each symptom is graduated from zero to five. This score classifies the symptoms of the lower urinary tract that will be assessed at randomization and after twelve months in each arm of the study.

SECONDARY OUTCOMES:
Occurrence of Acute Urinary Retention (AUR) | 12 months
  The occurrence of spontaneous obstruction of the urinary flow secondary to the benign prostatic hyperplasia.
Change from baseline Serum Creatinine | 12 months
  Serum creatinine values will be assessed at randomization and after twelve months
Change from baseline Serum Urea | 12 months
  Serum urea values will be assessed at randomization and after twelve months
Change from baseline Prostatic Specific Antigen (PSA) | 12 months
  Prostatic specific antigen serum values will be assessed at randomization and after twelve months.
Occurrence of Urinary infection | 12 months
  Occurrence of urinary tract infection during the study will be assessed through urine cultures
Adhesion to Medications | 12 months
  The adhesion to prescribed medications will be assessed after 12 months of the randomization

CONTACTS AND LOCATIONS:
Overall Officials: Brasil S Neto, MdPg, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital De Clinicas De Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carson C 3rd, Rittmaster R. The role of dihydrotestosterone in benign prostatic hyperplasia. Urology. 2003 Apr;61(4 Suppl 1):2-7. doi: 10.1016/s0090-4295(03)00045-1. PMID 12657354
- [Background] Davis DA, Thomson MA, Oxman AD, Haynes RB. Changing physician performance. A systematic review of the effect of continuing medical education strategies. JAMA. 1995 Sep 6;274(9):700-5. doi: 10.1001/jama.274.9.700. PMID 7650822
- [Background] Ferreira, J. B. B. et al. O complexo regulador da assistência à saúde na perspectiva de seus sujeitos operadores. Interface (Botucatu), Botucatu, v. 14, n. 33, June 2010
- [Background] Fratini, J. G.; Sauoe, R.; Massaroli, A. Referência e contra referência: contribuição para a integralidade em saúde. Cienc Cuid Saude, Itajaí, v. 7, n. 1, p. 65-72, Jan/Mar 2008
- [Background] Gusso, G.; Lopes, J. M. C. Tratado de Medicina de Família e Comunidade - 2 Volumes: Princípios, Formação e Prática. Artmed, 1ed., Porto Alegre, 2012
- [Background] Kirby RS. The natural history of benign prostatic hyperplasia: what have we learned in the last decade? Urology. 2000 Nov 1;56(5 Suppl 1):3-6. doi: 10.1016/s0090-4295(00)00747-0. PMID 11074195
- [Background] Mattos, L. A. P. et al. Desfechos clínicos aos 30 dias do registro brasileiro das síndromes coronárias agudas (ACCEPT). Arq. Bras. Cardiol., São Paulo, v.100, n. 1, Jan. 2013
- [Background] Platz EA, Smit E, Curhan GC, Nyberg LM, Giovannucci E. Prevalence of and racial/ethnic variation in lower urinary tract symptoms and noncancer prostate surgery in U.S. men. Urology. 2002 Jun;59(6):877-83. doi: 10.1016/s0090-4295(01)01673-9. PMID 12031373
- [Background] Starfield B. Primary care: an increasingly important contributor to effectiveness, equity, and efficiency of health services. SESPAS report 2012. Gac Sanit. 2012 Mar;26 Suppl 1:20-6. doi: 10.1016/j.gaceta.2011.10.009. Epub 2012 Jan 21. PMID 22265645
- [Background] Julious SA. Sample sizes for clinical trials with normal data. Stat Med. 2004 Jun 30;23(12):1921-86. doi: 10.1002/sim.1783. PMID 15195324
- [Background] Berger, Milton ; LUZ JR, Pedro Nery da ; SILVA NETO, Brasil ; KOFF, Walter José . Validação estatística do escore internacional de sintomas prostáticos (IPSS) na língua portuguesa. Jornal Brasileiro de Urologia, Rio de Janeiro/RJ, v. 25, n. 2, p. 225-234, 1999.
- See also: Portaria Ministério Da Saúde — http://bvsms.saude.gov.br/bvs/saudelegis/gm/2011/prt2546_27_10_2011.html